CLINICAL TRIAL: NCT00256659
Title: Hospital Outcomes: Intervention in Moderately III Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9808003482
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Moderately Ill Medical Inpatients at the Cornell Campus of the New York-Presbyterian Hospital
Keywords: Medical inpatients; Social Work; Physical therapy; Occupational therapy; Psychiatry; Early intervention; Iatrogenic complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Early assessment and referral to ancillary care services vs. standard care

SUMMARY:
To evaluate the utility of real time prognostic data (illness severity, stability and function) in the improvement of hospitalization morbidity, mortality, iatrogenic complications and length of stay.

DETAILED DESCRIPTION:
To evaluate resource allocation and efficiency of ancillary service delivery in aggregate cost and 3 month follow up in regards to hospital readmission, living environment, and utilization of social services.

This is a randomized study which will compare the current Standard of Care in hospital to EARLY assessment and referrals with respect to social work services, rehabilitation, psychiatry, and nursing. In this study, the control group will receive the hospital support services provided under current system of delivery and allocation. The intervention group will not receive any new or different services not already provided to all patients at New York Presbyterian Hospital. The difference between the 2 groups will be the uniformity of screening to identify the needs of the patient in the respective area of social services, rehabilitation, psychiatric assistance, and nursing care, and the timeliness by which the referrals for support services will be placed.

Potential interventions: (In both control and experimental group)

1. Social work: Discharge planning (homecare, visiting nursing services, skilled nursing facility placement).
2. Rehabilitation: Physical Therapy (improve ADLs-activities of daily living).
3. Psychiatry: Diagnosis and Assistance in management of Depression.
4. Nursing: Prevention of in hospital falls and decubitus ulcer formation.

ELIGIBILITY:
Inclusion Criteria:

1. All medical in-patients who are coded moderately ill with fair to poor function in the SIGNOUT program will be asked to participate in our study.
2. Patients who are able to provide verbal consent for their participation will be enrolled.

Exclusion Criteria:

1. Any patient not coded in the SIGNOUT system as moderately ill with fair to poor function.
2. Patients who refuses not to participate in the study.
3. Patients who are unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444
Dates: Start 1998-09; Study Completion 1999-04

PRIMARY OUTCOMES:
To evaluate the utility of real time prognostic data and in the improvement of hospitalization morbidity, mortality, iatrogenic complications, and length of stay.

SECONDARY OUTCOMES:
To evaluate resource allocation and efficiency of ancillary service delivery in aggregate cost and 3 month follow up in regards to hospital readmission, living environment, and utilization of social services.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University; James Hollenberg, MD, Principal Investigator — Weill Medical College of Cornell University; Mark Pecker, MD, Principal Investigator — Weill Medical College of Cornell University; Sona Euster, MSW, Principal Investigator — Weill Medical Center of Cornell University; Delia Gorga, PhD, Principal Investigator — Weill Medical Center of Cornell University; Mary Cooper, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital- Weill Medical Center, New York, New York, United States